CLINICAL TRIAL: NCT02375256
Title: A Phase I, Double-Blind, Randomized, Placebo-controlled Leukapheresis Study to Obtain Lymphocytes for the Study of Immune Responses in Healthy Adult Volunteers in the U.S. Who Receive BCG Vaccination Followed by Boosting With AERAS-402
Brief Title: A Leukapheresis Study for Immune Responses in Healthy US Adults Who Receive BCG Vaccination Followed by Boosting With AERAS-402
Acronym: C-021-402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-021-402
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — AERAS-402

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AERAS-402 (Experimental): 3 x10^10 viral particles per 0.5 mL suspended in 10 mM Tris buffer, 1 mM MgCl2, 75 mM NaCl, 5% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80), 0.1 mM EDTA, 10 mM l-histidine, 0.5% v/v ethanol and water. The dose volume administered was 0.5 mL.
  Interventions: Biological: AERAS-402; Biological: BCG (1-8 x105 cfu ID)
- Placebo (Active Comparator): 1.0 mL sterile vaccine buffer containing 10mM Tris buffer, 1 mM MgCl2, 75 mM NaCl, 5% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80), 0.1 mM EDTA, 10 mM l-histidine, 0.5% v/v ethanol and water. The dose volume administered was 0.5 mL
  Interventions: Biological: Placebo; Biological: BCG (1-8 x105 cfu ID)

INTERVENTIONS:
Biological: AERAS-402 — Live recombinant serotype 35 replication deficient adenovirus vector expressing a fusion protein of 3 Mycobacterium tuberculosis antigens (Ag85A, Ag85B, and TB10.4).
  Arms: AERAS-402
Biological: Placebo — Identical buffer solution in which AERAS-402 is formulated.
  Arms: Placebo
Biological: BCG (1-8 x105 cfu ID) — BCG given to all participants at day -84 prior to a boost with either Aeras-402 or placebo.

SUMMARY:
Healthy adults received BCG on Study Day -84, followed by randomization on Study Day 0 to receive 2 booster doses in a blinded fashion of either AERAS-402 (N=9) or placebo (N=2) on Study Days 0 and 28. Subjects were followed for a total of 98 days.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled study. At least 13, but no more than 16, subjects who met all eligibility criteria were to receive a prime vaccination with BCG (1-8 x 105 colony forming units [CFU] intradermally [ID]) at Study Day -84. Thirteen of the BCG-vaccinated subjects who completed all protocol-specified procedures and continued to meet eligibility criteria were to be enrolled and randomized on Study Day 0 in a 10:3 ratio to receive study vaccine (either AERAS-402 3 x 1010 virus particles [vp] intramuscularly [IM] or placebo IM) at Study Days 0 and 28, based on time of completion of screening. Eleven subjects were randomized (N=9 AERAS-402; N=2 placebo) and analyzed. Enrollment was stopped when 11 of the planned 13 subjects had been randomized, as it was felt that this number of subjects was sufficient to address the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female
2. Provided written informed consent prior to any study related procedures
3. Is age ≥18 years and ≤45 years on Study Day -84.
4. Has Body Mass Index (BMI) ≥19 and <33 by nomogram (see appendices)
5. Has general good health, confirmed by medical history and physical examination
6. Females physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must avoid pregnancy with an acceptable method of avoiding pregnancy from 28 days prior to Study Day -84 through the end of the study.
7. Females physically capable of pregnancy must have a negative serum pregnancy test within 7 days prior to Study Day -84 AND a negative urine pregnancy test on Study Day -84, Study Day 0, and Study Day 28.
8. Has committed to avoid elective surgery for the duration of the study
9. Has ability to complete all study visits as required per the protocol and is able to be contacted by telephone

Exclusion Criteria:

1. Acute illness, oral temperature ≥37.5°C, or axillary lymphadenopathy on Study Day -84, Study Day 0, or Study Day 28.
2. Any of the following laboratory results from blood and urine collected within 7 days prior to Study Day -84 (evaluated per local laboratory parameters):

   * Abnormal hemoglobin or hematocrit
   * Abnormal white blood cell count, absolute neutrophil count, or absolute lymphocyte count
   * Elevated creatinine, total bilirubin, AST, ALT, or alkaline phosphatase (ALP)
3. Evidence of chronic hepatitis (e.g., hepatitis B core antibody, or hepatitis C antibody, or other)
4. Laboratory test (e.g., QuantiFERON®-TB) evidence of Mycobacterium tuberculosis (Mtb) infection
5. History of residence in a tuberculosis-endemic country, per WHO 2008 "high-burden" definition
6. History of treatment for active or latent tuberculosis infection
7. History or evidence (including chest X-ray) of active tuberculosis
8. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
9. History of allergic disease or reactions likely to be exacerbated by any component of the BCG or study vaccines
10. History of autoimmune disease or immunosuppression
11. Current household contact or occupational exposure to an individual with known significant immunosuppression
12. History or evidence on physical examination of any systemic disease, or acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy
13. History or laboratory evidence of any past, present or future possible immunodeficiency state which will include (but is not limited to) any laboratory indication of HIV infection
14. History of alcohol or drug abuse within the past 2 years
15. History of cheloid formation
16. Previous medical history that may compromise the safety of the subject in the study
17. Any current medical, psychiatric, occupational, or substance abuse problems which, in the opinion of the investigator, will make it unlikely the subject will comply with the protocol
18. Inability to discontinue daily medications during the study period except the following:

    * Contraceptives
    * Multivitamins
    * Inhaled or topical corticosteroids
19. Tobacco smoking of a pack or more of cigarettes a day, or cannabis smoking three or more days per week
20. Received immunosuppressive medication within 45 days prior to Study Day -84 (inhaled and topical corticosteroids are permitted)
21. Received investigational drugs or vaccine products within 182 days prior to Study Day -84 or planned participation in any other investigational study during the study period
22. Received investigational Mtb vaccine at any time prior to Study Day -84
23. Received vaccination or immunotherapy with a BCG product at any time prior to Study Day -84.
24. Received immunoglobulin or blood products within 45 days prior to Study Day -84.
25. Received any standard vaccine within 45 days prior to Study Day -84 except inactivated influenza vaccine which may have been received within 2 weeks prior to Study Day -84.
26. History of high risk sexual behaviors since 1977.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cellular immune responses to AERAS-402 in healthy adult volunteers who received two booster doses of AERAS-402 administered 84 and 112 days after BCG vaccination, through leukapheresis and cryopreservation of cells followed by in vitro assay. | Up to study day 98
  percentage of CD4 and CD8 T cells from leukapheresis that produce any of three cytokines (IFN γ, TNF α, and/or IL 2).

SECONDARY OUTCOMES:
Evaluation of adverse events (AEs) and serious adverse events (SAEs). | Up to study day 98

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Ginsberg, MD PhD, Study Director — Aeras